CLINICAL TRIAL: NCT01177891
Title: Genetic Analysis of Familial Cases of Premature Ovarian Failure
Acronym: FAMIOP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM08084
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Familial Premature Ovarian Failure
MeSH Terms: conditions — Premature ovarian failure, familial

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Subject index: Population of familial cases of POF : 20 families with at least two subjects with POF nonsyndromic
- Population Index Related topics: Women, healthy women, men are potential carriers
- Population control: 100 Caucasian women with normal cycles until at least the age of 40 years and a proven fertility

SUMMARY:
The Premature ovarian failure (POF) is a rare syndrome observed in women under 40 who induced estrogen deficiency and often leads to infertility final. The etiologies of POF remain unknown in more than 85% of cases. There are 5-10 % of familial cases.The main objective of this study is to recruit, phenotype and genotype 20 families with at least two subjects with nonsyndromic POF in order to identify new loci using a single technical standard nucleotide polymorphisms (SNPs). This study will also include related population and population control.

DETAILED DESCRIPTION:
It was decided to move towards a study of familial cases of IOP. This study will identify areas of susceptibility in new families, identify candidate genes, sequence these genes in cases familial POF and sporadic cases in order to detect potential mutations, and in the control population.

ELIGIBILITY:
Inclusion Criteria:

Patients of familial cases of POF :

* Female subjects between 16 and 40 years or women older than 40 years with a cessation of ovarian function before the age of 40 years with increased levels of FSH
* Primary or secondary amenorrhea for more than three months with LH and FSH> 30mUI/ml
* No cases of fragile X syndrome in the family or blepharophimosis syndrome
* At least two cases in the family
* Origin Caucasian
* Patient signing the consent form for at least the blood sample
* Patient with Social Security

Population Index related topics :

* The presence of cycles until the age of 40 years with proven fertility, at least one child
* Amenorrhea and FSH> 30mUI/ml according to the criteria of the index subject
* Men of the family of index case

Population control :

* Women of Caucasian origin
* Women who had regular cycles until at least age 40 and at least one child
* Lack of land autoimmune (no history of thyroid disease or diabetes type 1)
* Woman signing the consent form for at least the blood sample

Exclusion Criteria:

* Blood donation of more than 450ml in the previous three months.
* Subject with an abnormal karyotype in favor of Turner syndrome or having a premutation of the FMR1 gene or a syndromic form
* Subject exclusion period in another study without direct individual benefit
* Subject refusing to sign the consent form

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Caucasian population
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Identification of candidate regions by genotyping within families | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Christin-Maitre, MD, PhD, Principal Investigator — Saint-Antoine hospital, Service of Endocrinology, ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS
Locations (2):
- France (2):
  - Hospital Saint-Antoine, Endocrinology service, Paris
  - Sophie Christin-Maitre, Paris

REFERENCES:
- [Background] Lebedin YS, Gorchakov VD, Petrova EN, Kobylyansky AG, Raudla LA, Tatarsky AR, Bobkov EV, Adamova IY, Vasilov RG, Nasonov EL, et al. Ex vivo removal of IgE in atopic asthma by extracorporeal plasmoimmunoadsorption (EPIA): development of a clinical adsorbent. Int J Artif Organs. 1991 Aug;14(8):508-14. PMID 1937940
- [Background] Knauff EA, Franke L, van Es MA, van den Berg LH, van der Schouw YT, Laven JS, Lambalk CB, Hoek A, Goverde AJ, Christin-Maitre S, Hsueh AJ, Wijmenga C, Fauser BC; Dutch POF Consortium. Genome-wide association study in premature ovarian failure patients suggests ADAMTS19 as a possible candidate gene. Hum Reprod. 2009 Sep;24(9):2372-8. doi: 10.1093/humrep/dep197. Epub 2009 Jun 9. PMID 19508998
- [Background] Charbit B, Christin-Maitre S, Demolis JL, Soustre E, Young J, Funck-Brentano C. Effects of testosterone on ventricular repolarization in hypogonadic men. Am J Cardiol. 2009 Mar 15;103(6):887-90. doi: 10.1016/j.amjcard.2008.11.041. Epub 2009 Jan 24. PMID 19268751
- [Background] Rousseau A, Ayoubi F, Deveaux C, Charbit B, Delmau C, Christin-Maitre S, Jaillon P, Uzan G, Simon T. Impact of age and gender interaction on circulating endothelial progenitor cells in healthy subjects. Fertil Steril. 2010 Feb;93(3):843-6. doi: 10.1016/j.fertnstert.2008.10.062. Epub 2008 Dec 25. PMID 19111297
- [Background] Warcoin M, Lespinasse J, Despouy G, Dubois d'Enghien C, Lauge A, Portnoi MF, Christin-Maitre S, Stoppa-Lyonnet D, Stern MH. Fertility defects revealing germline biallelic nonsense NBN mutations. Hum Mutat. 2009 Mar;30(3):424-30. doi: 10.1002/humu.20904. PMID 19105185
- [Background] Madelenat P, Koskas M; Groupe de reflexion sur la contraception progestative. [Update on the progestin-only contraception]. J Gynecol Obstet Biol Reprod (Paris). 2008 Nov;37(7):637-60. doi: 10.1016/j.jgyn.2008.06.013. Epub 2008 Sep 27. French. PMID 18824306
- [Background] Beysen D, De Jaegere S, Amor D, Bouchard P, Christin-Maitre S, Fellous M, Touraine P, Grix AW, Hennekam R, Meire F, Oyen N, Wilson LC, Barel D, Clayton-Smith J, de Ravel T, Decock C, Delbeke P, Ensenauer R, Ebinger F, Gillessen-Kaesbach G, Hendriks Y, Kimonis V, Laframboise R, Laissue P, Leppig K, Leroy BP, Miller DT, Mowat D, Neumann L, Plomp A, Van Regemorter N, Wieczorek D, Veitia RA, De Paepe A, De Baere E. Identification of 34 novel and 56 known FOXL2 mutations in patients with Blepharophimosis syndrome. Hum Mutat. 2008 Nov;29(11):E205-19. doi: 10.1002/humu.20819. PMID 18642388
- [Background] Chakhtoura Z, Bachelot A, Samara-Boustani D, Ruiz JC, Donadille B, Dulon J, Christin-Maitre S, Bouvattier C, Raux-Demay MC, Bouchard P, Carel JC, Leger J, Kuttenn F, Polak M, Touraine P; Centre des Maladies Endocriniennes Rares de la Croissance and Association Surrenales. Impact of total cumulative glucocorticoid dose on bone mineral density in patients with 21-hydroxylase deficiency. Eur J Endocrinol. 2008 Jun;158(6):879-87. doi: 10.1530/EJE-07-0887. Epub 2008 Apr 7. PMID 18390993
- [Background] Christin-Maitre S. [Physiology of ovulation and mode of action of contraceptive pills]. Rev Prat. 2008 Jan 15;58(1):17-20. French. PMID 18326357
- [Background] Christin-Maitre S. The role of hormone replacement therapy in the management of premature ovarian failure. Nat Clin Pract Endocrinol Metab. 2008 Feb;4(2):60-1. doi: 10.1038/ncpendmet0699. Epub 2007 Nov 20. No abstract available. PMID 18030288
- [Background] Tachdjian G, Aboura A, Portnoi MF, Pasquier M, Bourcigaux N, Simon T, Rousseau G, Finkel L, Benkhalifa M, Christin-Maitre S. Cryptic Xp duplication including the SHOX gene in a woman with 46,X, del(X)(q21.31) and premature ovarian failure. Hum Reprod. 2008 Jan;23(1):222-6. doi: 10.1093/humrep/dem358. Epub 2007 Nov 1. PMID 17981816
- [Background] Vinci G, Christin-Maitre S, Pasquier M, Bouchard P, Fellous M, Veitia RA. FOXO3a variants in patients with premature ovarian failure. Clin Endocrinol (Oxf). 2008 Mar;68(3):495-7. doi: 10.1111/j.1365-2265.2007.03052.x. Epub 2007 Sep 19. No abstract available. PMID 17888023
- [Background] Laissue P, Christin-Maitre S, Bouchard P, Fellous M, Veitia RA. Mutations in the NOG gene are not a common cause of nonsyndromic premature ovarian failure. Clin Endocrinol (Oxf). 2007 Jun;66(6):900. doi: 10.1111/j.1365-2265.2007.02797.x. Epub 2007 Mar 23. No abstract available. PMID 17381491
- [Background] Zanotti-Fregonara P, Khoury A, Duron F, Keller I, Christin-Maitre S, Kiffel T, Toubert ME, Devaux JY, Hindie E. Which thyroid cancer patients need periodic stimulation tests? Eur J Nucl Med Mol Imaging. 2007 Apr;34(4):541-6. doi: 10.1007/s00259-006-0279-z. Epub 2006 Nov 14. PMID 17106700
- [Background] Roux C, Briot K, Dumarcet N, Bourgoin M, Chapurlat R, Christin-Maitre S, Cortet B, Costagliola D, Diebolt V, Lacoin F, Letombe B, Oberlin F, Orcel P, Ravaud P, Seret P, Thomas T, Vogel JY, Barna A, Nouyrigat E, Veyries ML, Yoldjian I. [Drug treatment of postmenopausal osteoporosis. What's New in 2006]. Presse Med. 2006 Oct;35(10 Pt 2):1529-39. doi: 10.1016/s0755-4982(06)74847-3. No abstract available. French. PMID 17028517
- [Background] Laissue P, Christin-Maitre S, Touraine P, Kuttenn F, Ritvos O, Aittomaki K, Bourcigaux N, Jacquesson L, Bouchard P, Frydman R, Dewailly D, Reyss AC, Jeffery L, Bachelot A, Massin N, Fellous M, Veitia RA. Mutations and sequence variants in GDF9 and BMP15 in patients with premature ovarian failure. Eur J Endocrinol. 2006 May;154(5):739-44. doi: 10.1530/eje.1.02135. PMID 16645022
- [Background] De Baere E, Copelli S, Caburet S, Laissue P, Beysen D, Christin-Maitre S, Bouchard P, Veitia R, Fellous M. Premature ovarian failure and forkhead transcription factor FOXL2: blepharophimosis-ptosis-epicanthus inversus syndrome and ovarian dysfunction. Pediatr Endocrinol Rev. 2005 Jun;2(4):653-60. PMID 16208278
- [Background] Christin-Maitre S, Duron F. Fetal loss associated with excess thyroid hormone exposure. JAMA. 2004 Nov 3;292(17):2085-6; author reply 2086. doi: 10.1001/jama.292.17.2085-b. No abstract available. PMID 15523067
- [Background] Ouzounian S, Christin-Maitre S. [What is menopause?]. Rev Prat. 2005 Feb 28;55(4):363-8. French. PMID 15828613
- [Background] Simon T, Boutouyrie P, Gompel A, Christin-Maitre S, Laurent S, Thuillez C, Zannad F, Bernaud C, Jaillon P; CASHMERE investigators. Rationale, design and methods of the CASHMERE study. Fundam Clin Pharmacol. 2004 Feb;18(1):131-8. doi: 10.1111/j.1472-8206.2003.00233.x. PMID 14748765
- [Background] Hulot JS, Demolis JL, Riviere R, Strabach S, Christin-Maitre S, Funck-Brentano C. Influence of endogenous oestrogens on QT interval duration. Eur Heart J. 2003 Sep;24(18):1663-7. doi: 10.1016/s0195-668x(03)00436-6. PMID 14499229
- [Background] Christin-Maitre S, Ronci-Chaix N, Bouchard P. [Ovary genes and molecular pathology]. J Soc Biol. 2002;196(3):207-16. French. PMID 12462074
- [Derived] Rouen A, Rogers E, Kerlan V, Delemer B, Catteau-Jonard S, Reznik Y, Gompel A, Cedrin I, Guedj AM, Grouthier V, Brue T, Pienkowski C, Bachelot A, Chantot-Bastaraud S, Rousseau A, Simon T, Kott E, Siffroi JP, Touraine P, Christin-Maitre S. Whole exome sequencing in a cohort of familial premature ovarian insufficiency cases reveals a broad array of pathogenic or likely pathogenic variants in 50% of families. Fertil Steril. 2022 Apr;117(4):843-853. doi: 10.1016/j.fertnstert.2021.12.023. Epub 2022 Jan 31. PMID 35115167